CLINICAL TRIAL: NCT05083481
Title: A Phase 1/2 Study of ASP1570 as Monotherapy and in Combination With Pembrolizumab and/or Standard Therapies Including Chemotherapy and/or Immunotherapy in Participants With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of ASP1570 Taken by Itself, or ASP1570 Taken Together With Either Pembrolizumab, Standard Therapies, or Both, in Adults With Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1570-CL-0101; jRCT2031220527 (Registry Identifier: jRCT); KEYNOTE-E59 (Other: Merck Sharp & Dohme LLC); CTR20240514 (Registry Identifier: chinadrugtrials.org.cn); MK-3475-E59 (Other: Merck Sharp & Dohme LLC); 2023-505084-37 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-09-16; First posted 2021-10-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; ASP1570; Pembrolizumab
MeSH Terms: interventions — ASP1570; pembrolizumab; trifluridine tipiracil drug combination; Bevacizumab; Docetaxel; Oxaliplatin; Leucovorin; Fluorouracil; Irinotecan; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- ASP1570 Monotherapy Dose Escalation (Part 1) (Experimental): Participants will receive daily dose of ASP1570 in a 21-day cycle.
  Interventions: Drug: ASP1570
- ASP1570 + pembrolizumab Combination therapy Dose Escalation (Part 1) (Experimental): Participants will receive daily dose of ASP1570 in a 21-day cycle. pembrolizumab will be administered every 6 weeks on day 1 of every other ASP1570 cycle.
  Interventions: Drug: ASP1570; Drug: pembrolizumab
- ASP1570 + Docetaxel Combination therapy Dose Expansion - NSCLC 2L+ (Part 2) (Experimental): Participants who have NSCLC will receive RP2D of ASP1570 daily in a 21-day cycle. Docetaxel will be administered every 6 weeks on day 1 of every other ASP1570 cycle.
  Interventions: Drug: ASP1570; Drug: Docetaxel
- ASP1570 Monotherapy Dose Expansion - Food Effect (Part 2) (Experimental): Participants will receive RP2D of ASP1570 after the meal in a 21-day cycle. This cohort will be opened at the discretion of the sponsor.
  Interventions: Drug: ASP1570
- ASP1570 Monotherapy Dose Expansion - Intermittent dosing (Part 2) (Experimental): Participants will receive RP2D of ASP1570 with some periodical drug holiday in a 21-day cycle. This cohort will be opened at the discretion of the sponsor.
  Interventions: Drug: ASP1570
- ASP1570 Monotherapy Dose Expansion - Stepwise dosing (Part 2) (Experimental): Participants will receive ASP1570 administered by intra-subject dose escalation with gradual multiple dose steps (e.g., 3 steps) and increased dose up to RP2D in a 21-day cycle. This cohort will be opened at the discretion of the sponsor.
  Interventions: Drug: ASP1570
- ASP1570 Monotherapy Dose Expansion Microsatellite stable - colorectal cancer (MSS-CRC) (Part 2) (Experimental): Participants who have MSS-CRC will receive ASP1570 in a 21-day cycle.
  Interventions: Drug: ASP1570
- ASP1570 + TAS-102 + Bevacizumab Combination therapy Dose Expansion - MSS-CRC 3L+ (Part 2) (Experimental): Participants who have MSS-CRC will receive ASP1570 daily in a 28-day cycle. TAS-102 (Trifluridine + Tipiracil) will be administered on days 1 through 5 and days 8 through 12 of each 28-day cycle. Bevacizumab will be administered every 2 weeks.
  Interventions: Drug: ASP1570; Drug: Trifluridine + Tipiracil; Drug: Bevacizumab
- ASP1570 Monotherapy Dose Expansion NSCLC (Part 2) (Experimental): Participants who have NSCLC will receive ASP1570 in a 21-day cycle.
  Interventions: Drug: ASP1570
- ASP1570 + Pembrolizumab + Pemetrexed + Carboplatin CTDE - NSCLC 1L (Part 2) (Experimental): Participants who have NSCLC will receive ASP1570 daily in a 21-day cycle. Pembrolizumab will be administered every 6 weeks on day 1 of every other ASP1570 cycle. Pemetrexed and carboplatin will be administered on day 1 of each 21-day cycle.
  Combination therapy Dose Expansion (CTDE)
  Interventions: Drug: ASP1570; Drug: pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin
- ASP1570 + Bevacizumab + mFOLFOX6 or FOLFIRI Combination therapy Dose Expansion - MSS-CRC 2L (Part 2) (Experimental): Participants who have MSS-CRC will receive ASP1570 in a 14-day cycle. Bevacizumab, will be administered every 2 weeks. mFOLFOX6 (oxaliplatin, Leucovorin, 5-fluorouracil) or FOLFIRI (Leucovorin, 5-Fluorouracil, Irinotecan) will administered every 2 weeks.
  Interventions: Drug: ASP1570; Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-Fluorouracil; Drug: Irinotecan

INTERVENTIONS:
Drug: ASP1570 — Oral tablet
Drug: pembrolizumab — Intravenous Infusion
  Other Names: KEYTRUDA®
  Arms: ASP1570 + Pembrolizumab + Pemetrexed + Carboplatin CTDE - NSCLC 1L (Part 2); ASP1570 + pembrolizumab Combination therapy Dose Escalation (Part 1)
Drug: Trifluridine + Tipiracil — Oral Administration
  Other Names: TAS-102
  Arms: ASP1570 + TAS-102 + Bevacizumab Combination therapy Dose Expansion - MSS-CRC 3L+ (Part 2)
Drug: Bevacizumab — Intravenous Infusion
  Arms: ASP1570 + Bevacizumab + mFOLFOX6 or FOLFIRI Combination therapy Dose Expansion - MSS-CRC 2L (Part 2); ASP1570 + TAS-102 + Bevacizumab Combination therapy Dose Expansion - MSS-CRC 3L+ (Part 2)
Drug: Docetaxel — Intravenous Infusion
  Arms: ASP1570 + Docetaxel Combination therapy Dose Expansion - NSCLC 2L+ (Part 2)
Drug: Oxaliplatin — Intravenous Infusion
  Arms: ASP1570 + Bevacizumab + mFOLFOX6 or FOLFIRI Combination therapy Dose Expansion - MSS-CRC 2L (Part 2)
Drug: Leucovorin — Intravenous Infusion
  Arms: ASP1570 + Bevacizumab + mFOLFOX6 or FOLFIRI Combination therapy Dose Expansion - MSS-CRC 2L (Part 2)
Drug: 5-Fluorouracil — Intravenous Infusion
  Arms: ASP1570 + Bevacizumab + mFOLFOX6 or FOLFIRI Combination therapy Dose Expansion - MSS-CRC 2L (Part 2)
Drug: Irinotecan — Intravenous Infusion
  Arms: ASP1570 + Bevacizumab + mFOLFOX6 or FOLFIRI Combination therapy Dose Expansion - MSS-CRC 2L (Part 2)
Drug: Pemetrexed — Intravenous Infusion
  Arms: ASP1570 + Pembrolizumab + Pemetrexed + Carboplatin CTDE - NSCLC 1L (Part 2)
Drug: Carboplatin — Intravenous Infusion
  Arms: ASP1570 + Pembrolizumab + Pemetrexed + Carboplatin CTDE - NSCLC 1L (Part 2)

SUMMARY:
Immune therapies work with the body's immune system to treat a number of cancers. They work with T-cells, a type of white blood cell, to target and attack specific tumors. However, some tumors can become resistant to attack by T-cells over time. They do this by sending "off" signals to T-cells. The researchers are finding ways to switch the T-cells back on.

Before a treatment can be approved for use, clinical studies need to be done. This study will provide more information on ASP1570 in adults with advanced solid tumors. ASP1570 will either be given by itself, or given with another medicine called pembrolizumab, given with a standard cancer therapy, or given together with pembrolizumab and other medicines called pemetrexed and carboplatin.

The main aims of this study are：

* To check the safety of ASP1570
* To check how well ASP1570 is tolerated
* To find a suitable dose of ASP1570

This study is for adults with advanced solid tumors. Their tumor has either grown outside of the area where it started (locally advanced and unresectable) or it has spread to other parts of the body (metastatic). Their cancer gets worse after standard therapy or they are unable to have standard therapy. The study doctors can give more advice about who can take part.

This study will be in 2 parts.

In Part 1, the most suitable dose of ASP1570 to give to people with advanced solid tumors will be worked out. Different small groups of people with advanced solid tumors will take lower to higher doses of ASP1570. People will either be given ASP1570 by itself, or ASP1570 with pembrolizumab, ASP1570 with a standard cancer therapy, or ASP1570 with pembrolizumab, pemetrexed and carboplatin. The study treatment given depends on the type of cancer people have. There are different doses of ASP1570, with each group staying on the same dose. There is just 1 standard dose of pembrolizumab. The dose of a standard cancer therapy depends on its label. After taking the lowest dose of ASP1570, the first group will be checked for medical problems. The next group can only take the higher dose of ASP1570 if the first group tolerates the lowest dose. This will continue in the same way for each group.

Each group will take tablets of ASP1570 either once or twice every day in a 21-day cycle. People will continue with more treatment cycles on the same dose unless they can't tolerate the study treatment, their cancer gets worse or the study doctor decides that person should stop treatment. People who also receive treatment with pembrolizumab will be infused with pembrolizumab on the first day of every other cycle of ASP1570 (once every 6 weeks). People who are receiving a standard cancer therapy (with ASP1570) will be treated according to its label.

In Part 2, different small groups of people with advanced solid tumors will take the most suitable dose of ASP1570 worked out from Part 1. The dose will not go above the highest dose that people could tolerate from Part 1. ASP1570 will be given either once a day or twice a day in a 21-day cycle. Pembrolizumab will be given once every 6 weeks. Other study treatments will be given in 14-day, 21-day or 28-day cycles. The cycle length and other study treatments given (pembrolizumab and the type of standard cancer therapy will depend on what type of tumor people have. The standard cancer therapies will be given according to their label. All groups will continue with more treatment cycles with ASP1570 (by itself with pembrolizumab, with a standard cancer therapy, or with pembrolizumab, pemetrexed and carboplatin) unless they can't tolerate the study treatment, their cancer gets worse or the study doctor decides that person should stop treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant has locally-advanced (unresectable) or metastatic solid tumor malignancy which is confirmed by available pathology records or current biopsy.
* Participant has at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Monotherapy Escalation Cohorts and China-specific Safety Lead-in Cohort:

  a) Participant has progressed on standard therapies, is no longer eligible for standard therapies or has refused standard approved therapies (no limit to the number of prior treatment regimens). (UNIQUE to China: Certain tumor types with specific criteria may be prioritized at the sponsor's discretion).
* Monotherapy Expansion Cohorts:

  a) Participant has MSS-CRC or NSCLC and has progressed was intolerant to at least 2 prior anti-cancer therapy regimens administered for metastatic disease.
* Monotherapy Dose Optimization Cohorts:

  a) Participant has MSS-CRC or NSCLC and has progressed or was intolerant to at least 2 prior anti-cancer therapy regimens administered for metastatic disease.
* Combination Therapy Escalation and/or Expansion Cohorts:

  a) For NSCLC (2L+) Combination Therapy Cohort only:
* Participant has Stage IV NSCLC and has progressed on or after checkpoint inhibitors with or without platinum-based chemotherapy.
* Participant is eligible to receive docetaxel. b) For MSS-CRC (3L+) Combination Therapy Cohorts only:
* Participant must have progressed or was intolerant to at least 2 prior anti-cancer therapy regimens administered for metastatic disease.
* Participant is eligible to receive TAS-102 and bevacizumab.
* All Comers Combination with Pembrolizumab Cohorts only:
* Participant who has progressed on standard therapies, are no longer eligible for standard therapies or has refused standard approved therapies.
* Participant is eligible to receive pembrolizumab
* For NSCLC (1L) Combination Therapy Cohorts only:
* Participant has PD-L1 low (TPS = 1% to 49%) or negative (TPS < 1%) and AGA negative Stage IV adenocarcinoma (mixed histology is not allowed).
* Participant has not received prior systemic treatment for their advanced/metastatic NSCLC.
* Participant who remains disease free for 12 months following the completion of neoadjuvant/adjuvant treatment is eligible.
* Participant is eligible to receive pembrolizumab + pemetrexed + carboplatin.
* For MSS-CRC (2L) Combination Therapy Cohorts only:
* Participant is AGA negative and HER2 negative.
* mFOLFOX6 + Bevacizumab:
* Participant must have progressed or was intolerant to first line with irinotecan-based therapy, or previous therapy without oxaliplatin.
* Participant is eligible to receive mFOLFOX6 and bevacizumab.
* FOLFIRI + Bevacizumab:
* Participant must have progressed or was intolerant to first line with oxaliplatin-based therapy, or previous therapy without irinotecan.
* Participant is eligible to receive FOLFIRI and bevacizumab.
* Eligibility of backfill participants should follow cohort specific criteria for which they are being utilized.
* Participant has an Eastern Cooperative Oncology Group (ECOG) Status of 0 or 1 within 7 days before the first dose of study drug.
* Participant's adverse events (excluding alopecia) from prior anti-cancer therapies have resolved or improved to grade 1 at least 14 days prior to the first dose of study intervention. Note: Participants with type 1 diabetes mellitus and endocrinopathies stably maintained on appropriate replacement therapy are allowed.
* Participant has adequate organ function prior to start of study treatment (within 7 days prior to study intervention treatment initiation) as indicated by the following laboratory values. If a participant has received a recent blood transfusion, the laboratory tests must be obtained >= 2 weeks after any blood transfusion: Absolute Neutrophil Count (ANC) >= 1500/µL; Platelets >= 100,000/µL; Hemoglobin >= 9 g/dL (Criterion must be met without packed red blood cell transfusion within the 2 weeks prior. Participants can be on stable dose of erythropoietin (approximately ≥ 3 months); Creatinine clearance >= 45 mL/min (calculated by Cockcroft-Gault equation); Total Bilirubin either (a) <= 1.5 x ULN or (b) Direct bilirubin <= ULN and total bilirubin < 3 x ULN (for participants with Gilbert's syndrome); aspartate aminotransferase (AST) [serum glutamic oxaloacetic transaminase (SGOT)] and alanine aminotransferase (ALT) [serum glutamic pyruvic transaminase (SGPT)] <= 2.5 x ULN without liver metastases (or <= 5 x ULN if liver metastases are present); serum potassium >= 3.4mEg/L; serum magnesium >= 1.7mg/dL; serum ionized calcium >= 4.7 mg/dL; Thyroid stimulating hormone (TSH) within normal limits. Note: if TSH is not within normal limits at baseline, participant may still be eligible if T3 /or FT4 is within the normal limits.
* Participant has activated partial thromboplastin time and international normalized ratio (INR) <= 1.5 x ULN and is not receiving anticoagulation.
* Female participant is not pregnant confirmed by pregnancy test or confirmed to be of non-childbearing potential and at least one of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 45 days after final ASP1570 administration or at least 120 days after administration of pembrolizumab.
* Females participating in the study should be advised to use a highly effective contraception method during treatment and for 2 months after the last dose of docetaxel, and for 6 months after the last dose of TAS-102 and bevacizumab.
* Females participating in the study should be advised to use a highly effective contraception method during treatment and for 9 months after the last dose of mFOLFOX6.
* (UNIQUE to South Korea): Females participating in the study should be advised to use a highly effective contraception method during treatment and for 15 months after the last dose of mFOLFOX6.
* Females participating in the study should be advised to use a highly effective contraception method during treatment and for 6 months after the last dose of FOLFIRI.
* (UNIQUE to South Korea): Females participating in the study should be advised to use a highly effective contraception method during treatment and for 7 months after the last dose of FOLFIRI.
* Females participating in the study should be advised to use a highly effective contraception method during treatment and for 6 months after treatment with carboplatin, pemetrexed and pembrolizumab.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for at least 45 days after final ASP1570 administration or at least 120 days after administration of pembrolizumab.
* Females participating in the study should be advised to not breastfeed during and for 45 days after treatment of docetaxel.
* Females participating in the study should be advised to not breastfeed during treatment and for 6 months after the last dose of TAS-102 and bevacizumab.
* Females participating in the study should be advised to not breastfeed during treatment and for 45 days after the last dose of mFOLFOX6 or FOLFIRI.
* Females participating in the study should be advised to not breastfeed during treatment and for 4 months after treatment with a regimen of carboplatin, pemetrexed, and pembrolizumab.
* Female participant must not donate ova starting at first dose of study intervention and throughout the study period and for at least 45 days after final ASP1570 administration or at least 120 days after administration of pembrolizumab.
* Females participating in the study should be advised to not donate ova during treatment and for 2 months after the last dose of docetaxel.
* Females participating in the study should be advised to not donate ova during treatment and for 6 months after the last dose of TAS-102, bevacizumab or FOLFIRI.
* (UNIQUE to South Korea): Females participating in the study should be advised to not donate ova during treatment and for 7 months after the last dose of FOLFIRI.
* Females participating in the study should be advised to not donate ova during treatment and for 9 months after the last dose of mFOLFOX6.
* (UNIQUE to South Korea): Females participating in the study should be advised to not donate ova during treatment and for 15 months after the last dose of mFOLFOX6.
* Females participating in the study should be advised to not donate ova for 6 months after treatment with a regimen of carboplatin, pemetrexed and pembrolizumab.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for at least 45 days after final ASP1570 administration or at least 120 days after administration of pembrolizumab.
* Males participating in the study should be advised to use a highly effective contraception method during treatment and for 4 months after the last dose of docetaxel.
* Males participating in the study should be advised to use a highly effective contraception method during treatment and for 3 months after the last dose of TAS-102 and bevacizumab.
* Males participating in the study should be advised to use a highly effective contraception method during treatment and for 6 months after the last dose of mFOLFOX6.
* (UNIQUE to South Korea): Males participating in the study should be advised to use a highly effective contraception method during treatment and for 12 months after the last dose of mFOLFOX6.
* Males participating in the study should be advised to use a highly effective contraception method during treatment and for 3 months after the last dose of FOLFIRI.
* Males participating in the study should be advised to use a highly effective contraception method during treatment and for 6 months after the last dose of a regimen of carboplatin, pemetrexed and pembrolizumab.
* Male participant must not donate sperm during the treatment period and for at least 45 days after final ASP1570 administration or at least 120 days after administration of pembrolizumab.
* Males participating in the study must not donate sperm for at least 4 months after the last dose of docetaxel.
* Males participating in the study must not donate sperm for at least 3 months after the last dose of TAS-102 and bevacizumab.
* Males participating in the study must not donate sperm during treatment and for 6 months after the last dose of mFOLFOX6.
* (UNIQUE to South Korea): Males participating in the study should be advised to not donate sperm during treatment and for 12 months after the last dose of mFOLFOX6.
* Males participating in the study must not donate sperm during treatment and for 3 months after the last dose of FOLFIRI.
* Males participating in the study must not donate sperm during treatment and for 6 months after the last dose of a regimen of carboplatin, pemetrexed and pembrolizumab.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for at least 45 days after final ASP1570 administration or at least 120 days after administration of pembrolizumab.
* Males participating in the study with pregnant partner(s) should be advised to remain abstinent or use a condom during treatment and for 4 months after the last dose of docetaxel.
* Males participating in the study with pregnant partner(s) should be advised to remain abstinent or use a condom during treatment and for 6 months after the last dose of TAS-102 and bevacizumab.
* Males participating in the study with pregnant partner(s) should be advised to remain abstinent or use a condom during treatment and for 6 months after the last dose of mFOLFOX6.
* (UNIQUE to South Korea): Males participating in the study with pregnant partner(s) should be advised to remain abstinent or use a condom during treatment and for 12 months after the last dose of mFOLFOX6.
* Males participating in the study with pregnant partner(s) should be advised to remain abstinent or use a condom during treatment and for 3 months after the last dose of FOLFIRI.
* Males participating in the study with pregnant partner(s) should be advised to remain abstinent or use a condom during treatment and for 6 months after the last dose of a regimen of carboplatin, pemetrexed and pembrolizumab.
* Participant agrees not to participate in another interventional study while receiving study treatment in the present study.

Exclusion Criteria:

* Participant has received antineoplastic therapy, including investigational therapy within 28 days or 5 half-lives (whichever is shorter) (antitumor traditional Chinese medicine within 14 days) prior to the start of study intervention administration.
* Participant requires or has received systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to the first dose of IP. Participants using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 10 mg prednisone) are allowed.
* Participant requires strong or moderate CYP2D6 inhibitors (e.g., bupropion, fluoxetine, paroxetine, duloxetine, abiraterone) during the study.
* Participant has symptomatic central nervous system (CNS) metastases or participant has evidence of unstable CNS metastases even if asymptomatic (e.g., progression on scans). Participants with previously treated CNS metastases are eligible, if they are clinically stable and have no evidence of CNS progression by imaging for at least 4 weeks prior to start of study treatment and are on a stable dose of ≤ 10 mg/day of prednisone or equivalent for at least 2 weeks (if requiring steroid treatment). Participant does not have leptomeningeal disease.
* Participant has an autoimmune disease. Participants with type 1 diabetes mellitus, endocrinopathies stably maintained on appropriate replacement therapy are allowed.
* Participant was discontinued from prior immunomodulatory therapy due to a toxicity that requires permanent discontinuation per toxicity management guidelines that was mechanistically related (e.g., immune related) to the agent.
* Participant has a known history of human immunodeficiency virus (HIV) infection. However, participants with HIV with cluster of differentiation 4 (CD4)+ T-cell counts ≥ 350 cells/µL and no history of AIDS-defining opportunistic infections within the past 6 months are eligible. NOTE: Screening for HIV infection should be conducted per local requirements.
* Participant has any of the following per screening serology test:

  * Hepatitis A virus (HAV) antibodies (immunoglobulin M [IgM])
  * Positive hepatitis B surface antigen (HBsAg). For participants with negative HBsAg, but positive HBcAB, an HBV DNA test will be performed and if positive the participants will be excluded.
  * Hepatitis C virus (HCV) antibodies unless HCV RNA is undetectable
* Participant has received a live or live attenuated vaccine against infectious diseases within 28 days prior to the first dose of study intervention.
* Participant has a history of noninfectious pneumonitis/interstitial lung disease [ILD], that required steroids, or currently has pneumonitis/interstitial lung disease.
* Participant has received prior radiotherapy within 2 weeks of start of study treatment or have had a history of radiation pneumonitis.

Note: Participants must have recovered from all radiation-related toxicities and not require corticosteroids > 10 mg per day of prednisone or equivalent. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.

* Participant has an infection requiring systemic therapy within 14 days prior to the first dose of study intervention.
* Participant has received a prior allogenic hematopoietic stem cell transplant or solid organ transplant.
* Participant is expected to require another form of antineoplastic therapy while on study treatment.
* Participant has had a myocardial infarction or unstable angina within 6 months prior to the start of study treatment or currently has an uncontrolled illness including, but not limited to symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participant has inadequately controlled hypertension (defined as systolic blood pressure >= 140 and/or diastolic blood pressure >= 90 mmHg on antihypertensive medications, or systolic blood pressure > 130 and/or diastolic blood pressure > 80 mmHg without antihypertensive medications).
* Participant has a corrected QT interval using Fridericia's formula (QTcF) > 450 msec (for male and female participants) during screening. ECGs will be performed in triplicate during screening. (The average of the triplicate readings will be used in the calculation for corrected QT interval [QTc]).
* Participant has a prior malignancy, other than the current malignancy for which the participant is seeking treatment, active (i.e., requiring treatment or intervention) within the previous 2 years except for locally curable malignancies that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.
* Participant has had a major surgical procedure and has not completely recovered within 28 days prior to the first dose of study intervention.
* Participant has a history of bleeding diathesis that makes the participant unsuitable for study participation.
* Participant requires use of any anticoagulation therapy.
* Participant has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the participant to participate in the study.
* Participant has a known or suspected hypersensitivity to ASP1570. For participants entering combination therapy, they have a known or suspected hypersensitivity to the respective standard therapy study intervention (pembrolizumab, docetaxel, TAS 102, mFOLFOX6, FOLFIRI and/or bevacizumab), or any components of the formulation used.
* For the combination therapies, participant has received radiation therapy to the lung that is > 30 Gy within 6 months of the first dose of study intervention.
* All Solid Tumors Combination Therapy Cohort only: HIV-infected participants with a history of Kaposi sarcoma and/or multicentric Castleman disease.
* Dose escalation combination therapy, dose expansion combination therapy, dose expansion monotherapy, China safety lead in and backfill participants: participants with known actionable driver mutation (e.g., EGFR, ALK, NTRK).
* Previous therapy with DGK inhibitor is prohibited.
* Participants with a history of or ongoing sensory or motor neuropathy Grade 2 or higher.
* Participants with a history of ≥ Grade 2 hearing loss (only for NSCLC [1L] combination therapy cohort with carboplatin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) for ASP1570 Single Agent | 21 days
  A DLT is defined as any event meeting the DLT criteria occurring within 21 days of first dose on Cycle 1 Day 1 (C1D1), excluding toxicities clearly related to disease progression or intercurrent illness.
Number of Participants with Adverse Events (AEs) | Up to 27 months
  Adverse events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a participant temporally associated with the use of study IP, whether or not considered related to the study IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study IP. This includes events related to the comparator and events related to the (study) procedures.
Change from baseline to 45 days after End of Treatment (EOT) in laboratory values | Baseline and 45 days after EOT
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade changes from baseline to highest post-baseline grade will be assessed.
Number of participants with vital sign abnormalities and/or AEs | Up to 27 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to 24 months
  Number of participants with potentially clinically significant ECG values.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) of ASP1570 per Immune Response Evaluation Criteria in Solid Tumors (iRECIST) | Up to 27 months
  ORR is defined as the proportion of participants for each dose level whose best overall response is rated as Complete Response (CR) or Partial Response (PR) per iRECIST.
ORR of ASP1570 per Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1) | Up to 27 months
  ORR is defined as the proportion of participants for each dose level whose best overall response is rated as Complete Response (CR) or Partial Response (PR) per RECIST 1.1.
Duration of Response (DOR) of ASP1570 per iRECIST | Up to 27 months
  DOR will be calculated only for the subgroup of participants with confirmed response CR/PR per iRECIST.
Duration of Response (DOR) of ASP1570 per RECIST 1.1 | Up to 27 months
  DOR will be calculated only for the subgroup of participants with confirmed response CR/PR per RECIST 1.1.
Disease Control Rate (DCR) of ASP1570 per iRECIST | Up to 27 months
  DCR is defined as the proportion of participants for each dose level whose best overall response is rated as confirmed CR, PR or SD per iRECIST.
Disease Control Rate (DCR) of ASP1570 per RECIST 1.1 | Up to 27 months
  DCR is defined as the proportion of participants for each dose level whose best overall response is rated as confirmed CR, PR or SD per RECIST 1.1.
Pharmacokinetics of ASP1570 in plasma: Maximum Concentration (Cmax) | Up to 27 months
  Cmax will be recorded from the PK plasma samples collected.
Pharmacokinetics of ASP1570 in plasma: Time of Maximum Concentration (tmax) | Up to 27 months
  tmax will be recorded from the PK plasma samples collected.
Pharmacokinetics of ASP1570 in plasma: Area under the plasma concentration-time curve during a dosage interval (AUCtau) | Up to 27 months
  AUCtau will be recorded from the PK plasma samples collected.
Pharmacokinetics of ASP1570 in plasma: Trough plasma concentration (Ctrough) | Up to 27 months
  Ctrough will be recorded from the PK plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (43):
- United States (16):
  - Providence Medical Foundation, Fullerton, California
  - California Research Institute, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Florida Cancer Specialist & Research Institute Sarasota, Sarasota, Florida
  - University of Chicago, Chicago, Illinois
  - University of Kentucky Medical Center MCC-CRO, Lexington, Kentucky
  - American Oncology Partners, Bethesda, Maryland
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Atlantic Health System/Morristown Medical Center, Morristown, New Jersey
  - Columbia University, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Mary Crowley Research Center, Dallas, Texas
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
- China (5):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Second Affiliated Hospital Zhejiang University School of Medicine (SAHZU), Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Shanghai East Hospital, Shanghai
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
- France (7):
  - FR33007, Besançon
  - Site FR33002, Bordeaux
  - FR33008, Paris
  - FR33001, Poitiers
  - FR33005, Saint-Herblain
  - FR33009, Toulouse
  - Site FR33004, Villejuif
- Japan (6):
  - Aichi Cancer Center, Chikusa-ku, Nagoya-City, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital Of JFCR, Koto-ku, Tokyo
- Puerto Rico Medical Center, Río Piedras, Puerto Rico
- KR82002, Seoul, South Korea
- Spain (7):
  - Site ES34005, A Coruña, Barcelona
  - Site ES34004, Avda
  - Site ES34002, Madrid
  - ES34008, Málaga
  - Site ES34007, Málaga
  - Site ES34006, Pozuelo de Alarcón
  - ES34003, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/